CLINICAL TRIAL: NCT04723628
Title: The Effect of Telephone Consultancy Based on the Information, Motivation and Behavioral Skills Model on HbA1c and Self-Management for Individuals With Type 2 Diabetes: A Randomized Controlled Trial
Brief Title: The Effect of Telephone Consulting on HbA1 and Self-Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University (Other)
Responsible Party: Principal Investigator, KADRİYE SAYIN KASAR, PhD, RN, Aksaray University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AksarayU
Record Dates: First submitted 2021-01-18; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Type 2 Diabetes; Self-management
Keywords: Type 2 diabetes; Telephone counseling; IMB; Self-management; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Then, each patient was given 45-60 minutes of individual instruction. The patient training content was prepared based on the Knowledge, Motivation and Behavioral Skills Model (IMB). A total of 12 weeks of follow-up was performed with a weekly short reminder message and a two-weekly phone call. The research data were collected again at the end of 12 weeks.
  Interventions: Behavioral: Intervention group (telephone counseling)
- Control group (No Intervention): All data forms were then completed, and the HbA1c value was taken from the medical data. No additional procedure was performed to the control group. The research data were collected again at the end of 12 weeks.

INTERVENTIONS:
Behavioral: Intervention group (telephone counseling) — Then, each patient was given 45-60 minutes of individual instruction. The patient training content was prepared based on the Knowledge, Motivation and Behavioral Skills Model (IMB). A total of 12 weeks of follow-up was performed with a weekly short reminder message and a two-weekly phone call. The research data were collected again at the end of 12 weeks.
  Arms: Experimental group

SUMMARY:
The aim of this study was to investigate the effect of telephone counseling (12 weeks) based on the Information, Motivation, Behavioral Skills (IMB) Model in patients with type 2 diabetes mellitus (T2DM) on self-management and HbA1c.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effect of telephone counseling based on the Information, Motivation, Behavioral Skills (IMB) Model in patients with type 2 diabetes mellitus (T2DM) on self-management and HbA1c. This study was conducted with a randomized controlled trial. This study, between January 2019 and September 2019 were conducted in endocrine clinic. A total of 63 patients (31 interventions, 32 controls) diagnosed with T2DM were included. The intervention group received 45-60 minutes of patient training based on the Information, Motivation and Behavioral Skill Model (IMB). A weekly short reminder message and a two-weekly phone call were made and a total of 12 weeks of follow-up was conducted. As a result, there was a statistically significant difference between pre-test HbA1c, weight and systolic blood pressure (p<0.05). Also, after three months of follow-up, self-efficacy, self-management and self-management perceptions were significantly higher in the intervention group (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with type 2 DM at least six months previously
* Using a mobile phone
* HbA1c greater than 7%
* Living in the city
* Physical and mental health levels adequate for participation in the research

Exclusion Criteria:

* Having severe hearing or perceptual deficits that impaired communication
* Patients who did not agree to participate in the study
* Receiving inpatient treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Glycemic Control | 3 months
  Glycated hemoglobin (HbA1c) is the most widely used measure of glycemic control. A blood test was used to obtain HbA1c.

SECONDARY OUTCOMES:
Type 2 Diabetes Self-Efficacy Scale | 3 months
  The lowest score obtainable from the scale is 20, and the highest is 100. In the general evaluation of the scale according to the total mean score obtained based on the mean scores of all the subscales, those below the mean score are accepted as low self-efficacy and those above the mean score are accepted as high self-efficacy.
Diabetes Self-Management Questionnaire (DSMQ) | 3 months
  This scale is an individual assessment scale consisting of 16 items to investigate the relationship between diabetes self-management and diabetes control in glycemic control.
Perceived Diabetes Self-Management Scale (PDSMS) | 3 months
  The minimum score which can be obtained from the scale is 8 and the maximum score is 40. A higher total score obtained indicates a better awareness by the person of diabetes management.

CONTACTS AND LOCATIONS:
Locations (1):
- Kadriye Sayin Kasar, Aksaray, İlçe Seçiniz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sayin Kasar K, Duru Asiret G, Kutmec Yilmaz C, Canlar S. The effect of model-based telephone counseling on HbA1c and self-management for individuals with type 2 diabetes: A randomized controlled trial. Prim Care Diabetes. 2022 Feb;16(1):41-48. doi: 10.1016/j.pcd.2021.09.005. Epub 2021 Sep 11. PMID 34518109